CLINICAL TRIAL: NCT04492332
Title: Influencing Factors of Intracranial Hypertension in Patients With Bilateral Transverse Sinus Stenosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Ji Xunming,MD,PhD, Professor, Capital Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: BTSS-ICP
Record Dates: First submitted 2020-06-12; First posted 2020-07-30 (Actual); Last update posted 2020-07-30 (Actual); Status verified 2020-07

CONDITIONS: Vertebral Venous Collaterals; Serum Uric Acid; Intracranial Hypertension; Bilateral Transverse Sinus Stenosis
Keywords: vertebral venous collaterals; serum uric acid; Bilateral transverse sinus stenosis; intracranial hypertension
MeSH Terms: conditions — Intracranial Hypertension

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- normal controls with VVC (Sham Comparator): BTSS was confirmed by two of magnetic resonance venography (MRV), computed tomography venography (CTV) or digital subtraction angiography (DSA). The index of TSS (ITSS) score was a useful tool for the assessment of BTSS severity. The degree of stenosis was graded from 0 to 4 based on the following scale: 0 = normal; 1 = stenosis up to 1/3; 2 = stenosis between 1/3 and 2/3; 3 = stenosis >2/3; and 4 = hypoplasia. ITSS was calculated as degree of right TSS × degree of left TSS. Vertebral venous collaterals (VVC) were found.
  Interventions: Diagnostic Test: standard lumbar puncture
- normal controls without VVC (Sham Comparator): BTSS was confirmed by two of magnetic resonance venography (MRV), computed tomography venography (CTV) or digital subtraction angiography (DSA). The index of TSS (ITSS) score was a useful tool for the assessment of BTSS severity. The degree of stenosis was graded from 0 to 4 based on the following scale: 0 = normal; 1 = stenosis up to 1/3; 2 = stenosis between 1/3 and 2/3; 3 = stenosis >2/3; and 4 = hypoplasia. ITSS was calculated as degree of right TSS × degree of left TSS. Vertebral venous collaterals (VVC) were not found.
  Interventions: Diagnostic Test: standard lumbar puncture
- BTSS patients with VVC (Active Comparator): BTSS was confirmed by two of magnetic resonance venography (MRV), computed tomography venography (CTV) or digital subtraction angiography (DSA). The index of TSS (ITSS) score was a useful tool for the assessment of BTSS severity. The degree of stenosis was graded from 0 to 4 based on the following scale: 0 = normal; 1 = stenosis up to 1/3; 2 = stenosis between 1/3 and 2/3; 3 = stenosis >2/3; and 4 = hypoplasia. ITSS was calculated as degree of right TSS × degree of left TSS. Vertebral venous collaterals (VVC) were found.
  Interventions: Diagnostic Test: standard lumbar puncture
- BTSS patients without VVC (Active Comparator): BTSS was confirmed by two of magnetic resonance venography (MRV), computed tomography venography (CTV) or digital subtraction angiography (DSA). The index of TSS (ITSS) score was a useful tool for the assessment of BTSS severity. The degree of stenosis was graded from 0 to 4 based on the following scale: 0 = normal; 1 = stenosis up to 1/3; 2 = stenosis between 1/3 and 2/3; 3 = stenosis >2/3; and 4 = hypoplasia. ITSS was calculated as degree of right TSS × degree of left TSS. Vertebral venous collaterals (VVC) were not found.
  Interventions: Diagnostic Test: standard lumbar puncture

INTERVENTIONS:
Diagnostic Test: standard lumbar puncture — Subjects underwent a standard lumbar puncture to measure the intracranial pressure (ICP). ICP was measured invasively through lumbar space in the morning.

SUMMARY:
Bilateral transverse sinus stenosis (BTSS) is associated with intracranial hypertension (IH). However, not every BTSS patients presented with IH. The risk factors of IH in BTSS patients remained obscure. Vertebral venous collaterals (VVC) were often found in patients with bilateral transverse sinus stenosis (BTSS). The purpose of this study was to investigate the physiological role of VVC in BTSS patients.

DETAILED DESCRIPTION:
Bilateral transverse sinus stenosis (BTSS) is characterized by narrowing of bilateral transverse sinus which resulted in obstruction of venous reflux. The majority of BTSS patients exhibited with intracranial hypertension (IH) which manifested as a triad of headaches, tinnitus and papilledema. Stenting improved the symptoms in patients with transverse sinus stenosis (TSS) and reduced the elevated intracranial pressure (ICP). It is suggested that BTSS is one of the etiologies of IH. Since an alternative pattern of venous reflux was observed in patients with occluded superior sagittal sinus, it is postulated that altered pattern of venous reflux also exists in the presence of BTSS. The drainage of cerebral veins consists of two major pathways: transverse sinus-sigmoid sinus-internal jugular vein and vertebral venous plexus. Vertebral venous plexus is an extensive paravertebral system that provides direct venous communication between peritoneum and cranial cavity. The presence of vertebral venous collaterals (VVC) was reported in 108 consecutive patients. However, whether VVC is of physiological significance in BTSS patients remained unknown. This study was aimed to investigate the physiological role of VVC and whether it is involved in the regulation of IH and related clinical symptoms in BTSS patients.

Besides, it is presumed that serum uric acid (UA) may affect the formation of vertebral venous collaterals (VVC) and intracranial pressure (ICP). It is reported that UA inhibits the endothelial NO biological activity. High concentrations of uric acid (UA) suppresses circulating VEGF in Wistar rats and VEGF secretion in human endothelial cells. It is presumed that serum UA may affect the formation of VVC and ICP. The aim of this study is to investigate whether serum UA serves as an influencing factor of VVC and an indicator of IH in BTSS patients.

ELIGIBILITY:
Inclusion Criteria:

* BTSS confirmed by two of magnetic resonance venography (MRV), computed tomography venography (CTV) or digital subtraction angiography (DSA).

Exclusion Criteria:

* medicine related intracranial hypertension;
* systemic inflammation;
* moderate to severe stenosis in intracranial, carotid or vertebral arteries;
* moderate to severe stenosis in intracranial or jugular veins other than transverse sinus;
* intracranial lesions.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 137 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
intracranial pressure (ICP) | at admission
  ICP was detected by standard lumbar puncture

SECONDARY OUTCOMES:
serum uric acid (UA) | at admission
  Fasting venous blood was withdrawn simultaneously to assess serum UA.

OTHER OUTCOMES:
Triad of IH: papilledema | at admission
  Fundus photography was graded by using modified Frisén's grade
Triad of IH: headache | at admission
  10-point Numeric Pain Rating Scale (NPRS)
Triad of IH: tinnitus | at admission
  questionnaires for tinnitus handicap inventory (THI)

CONTACTS AND LOCATIONS:
Locations (1):
- Xuanwu Hospital, Beijing, China